CLINICAL TRIAL: NCT06976424
Title: Comparison of Eflornithine Cream Combined With Intense Pulsed Light Versus Intense Pulsed Light Alone for Hirsutism in Women
Brief Title: Comparison of a Face Cream Plus a Laser Procedure and Face Cream Alone in Treatment of Excessive Face Hairs in Female
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Umaima Nazar, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59/DME/KMC
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hirsuitism
Keywords: Hirsuitism; IPL; Eflornithine
MeSH Terms: conditions — Hirsutism | interventions — Eflornithine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupA (Experimental): This group is treated with combination of eflornithine cream and intense pulsed light for a period of three month.
  Interventions: Radiation: Instense pulsed light; Drug: Eflornithine Topical
- Group B (Experimental): This group is treated with eflornithine cream twice daily only for a period of three month
  Interventions: Drug: Eflornithine Topical

INTERVENTIONS:
Drug: Eflornithine Topical — Eflornithine cream will be applied to the face of group B female patients
  Other Names: Eflornithine cream
  Arms: Group B
Radiation: Instense pulsed light — Intense pulse light will be applied to the face of patient of Group A on areas having increase hair. Patient will be called for a followup every month for next session.
  Arms: GroupA
Drug: Eflornithine Topical — Eflornithine will be given to group A patient along with intense pulsed light and results will be compared to group B who recieved only Eflornithine cream
  Arms: GroupA

SUMMARY:
The study compares the effects of a cream alone and a combined effect of cream and laser for the treatment of excessive facial hairs in women .

DETAILED DESCRIPTION:
Hirsuitism refers to excessive terminal hairs in females, following a distribution pattern typically associated with male. It is associated with either increase response of hair follicles to androgen or either increase level of circulating androgens.The treatment options available are topical creams like eflornithine and laser treatments for hair removal. This study aims to conduct the comparison of a eflornithine cream and intense pulsed light laser versus eflornithine cream alone for the treatment of excessive facial hairs.

ELIGIBILITY:
Inclusion Criteria:

Gender (Female) Age between 18-45 Years Women with hirsutism as mentioned in the operational definition

Exclusion Criteria:

Pregnant women Women with severe acne Women with immunodeficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All the female patients with excessive facial hairs were included in the study.
Enrollment: 122 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment | 3 months
  Efficacy of treatment is defined as complete clearance of excessive hairs assesed on the basis of 4- level scale ranging 0 to 3 after 3 months of administration of the treatment in both groups.
  Clear is grade 3 Marked improvement is grade2 Improved is grade1 No improvement is grade 0

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Khyber Teaching Hospital, Peshawar, Kpk
  - Khyber Teaching Hospital, Peshawar, KPK
  - Khyber Teachinng Hospital, Peshawar, KPK

IPD SHARING:
Plan to Share IPD: No
Because the confedentiality of the patient would be breached.